CLINICAL TRIAL: NCT01440400
Title: The Use of Ultrasound to Guide Spinal Anesthesia in Obstetrics. Is There an Advantage Over Landmark Technique in Non-obese Patients?
Brief Title: Ultrasound Guided Spinal Anesthesia in Non Obese Obstetric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corniche Hospital (Other)
Responsible Party: Principal Investigator, Dr. Tarek Ansari, Consultant anesthetist, Corniche Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ch3151105
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Cesarean Section
Keywords: Ultrasound; Spinal anesthesia; Cesarean section

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional spinal anesthesia (No Intervention)
- Ultrasound guided spinal anesthesia (Experimental)
  Interventions: Procedure: Ultrasound guided spinal anesthesia

INTERVENTIONS:
Procedure: Ultrasound guided spinal anesthesia — Using the ultrasound to identify the spinal puncture level, mid-line and the depth of the dura.
  Arms: Ultrasound guided spinal anesthesia

SUMMARY:
The classical method for spinal anesthesia relies on the use of bony landmarks to identify the level and point of entry of the spinal needle. Over the years, in experienced hands, this method consistently proved to be successful and safe.

The introduction of ultrasound to guide neuraxial anaesthesia into clinical practice was relatively slow compared to peripheral nerve blocks or central venous catheterization. This could be due to the technical difficulties posed by the bony structures surrounding the spinal cord and its dura that blocks the path of the ultrasound beam. Many anesthetists are reluctant to change their conventional landmark technique, particularly with most studies showing no change in the success rate between ultrasound guided and the landmark techniques.

Several studies however showed that the ultrasound guided approach reduces the number of attempts to achieve a successful block and reduces the procedure time particularly in obese patients and those with technical difficulties.

In this study the investigators are trying to answer the following question : Is there any advantage in using ultrasound to guide spinal anaesthesia in non obese obstetric patients with easily palpable bony landmarks?

DETAILED DESCRIPTION:
Patients will be randomized using a web based randomization program into two groups: Ultrasound guided spinal anesthesia (US) & conventional spinal anesthesia (C). In both groups, the level of the third or fourth lumbar inter-space (L3/4 or L4/5) will be identified using either ultrasound (transverse and longitudinal approach) or palpation method using anatomical landmarks.

All ultrasound examinations and spinal anesthesia will be performed by 3 anesthetists with experience in ultrasound guided neuraxial block (between 100 and 200 cases). The ultrasound examination will be done using Logiq e TM ultrasound machine (GE Solingen Germany) with 4C RS 2 - 5.5MHz Broadband multi-frequency probe.

The predetermined point of entry for the introducer needle will be marked on the patient's back. The spinal anaesthesia will be administered with the patient in the sitting position, using a 26 gauge pencil point needle (PortexTM) with 15 mg of heavy Bupivacaine and 20 micrograms of Fentanyl. An independent observer, who is blinded to the method used to identify the point of entry of the introducer needle, will be collecting the data.The spinal anesthesia will be labeled as successful if a bilateral block to the sixth thoracic dermatome (T6) , judged by loss of cold and touch discrimination, is established 5 minutes after the spinal injection.

ELIGIBILITY:
Inclusion Criteria:

* All mothers with body mass index (BMI) equal to or less than 35 who has normal singleton pregnancy
* At 37 weeks gestation or more
* Admitted to Corniche Hospital for elective caesarean section under spinal anaesthesia

Exclusion Criteria:

* Patients with BMI >35
* Patieints with difficult anatomical landmarks
* Patients with neurological disease or coagulation defects
* Patients receiving anticoagulants
* Patients refusing spinal anaesthesia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The number of skin punctures | 30 minutes
  Number of times the skin is punctured by the introducer needle.
The number of spinal needle passes | 30 minutes
  The number of times the spinal needle tip is advanced beyond the tip of the introducer needle.
The time of the procedure | 30 minutes
  From skin puncture by the introducer to viewing cerebro-spinal fluid back-flow at the hub of the spinal needle.

SECONDARY OUTCOMES:
The patient satisfaction with spinal anesthesia | 24 hours
  scale 0-10, 0=not satisfied, 10=completely satisfied
Backache after spinal needle placement, assessed within 24 hours postoperatively | 24 hours
  verbal rating scale(VRS), 0-10, 0=no pain, 10=maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Ansari, FFARCSI, Principal Investigator — Corniche Hospital; Mounir Fayez, MD, Principal Investigator — Corniche Hospital; Amr Maher, MD, Principal Investigator — Corniche Hospital; Ahmed El Gamassy, MD, Principal Investigator — Corniche Hospital
Locations (1):
- Corniche hospital, Abu Dhabi, United Arab Emirates